CLINICAL TRIAL: NCT00234611
Title: Localization of CRT According to Echocardiography: LOCATE-Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Michigan Heart, PC (Other)
Collaborators: Medtronic (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MH-MDT-01
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2006-11-06 (Estimated); Status verified 2006-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Procedure: Echocardiogram guided left ventricular lead placement

SUMMARY:
Currently, the majority of heart failure patients who qualify for and receive a cardiac resynchronization therapy (CRT) device feel better than before their implant. However, there are some patients who do not improve after the implant. Michigan Heart is sponsoring a research study called LOCATE-Pilot to help understand whether the information from an echocardiogram, performed before implanting the CRT device, improves patients' responses to CRT. This is being done by evaluating your heart's function with an echocardiogram, to measure your heart's response during therapy. The study hypothesis is that response to CRT may be optimized by guiding left ventricular lead placement to the maximally delayed, viable basal segment of the left ventricle.

DETAILED DESCRIPTION:
CRT is a promising treatment modality for medically-refractory New York Heart Association (NYHA) class III or IV heart failure (HF) patients with intraventricular conduction delay (QRS > 130 ms). The randomized trials also suggest that a substantial minority of patients do not benefit, either echocardiographically or clinically, from CRT. In the MIRACLE trial, for instance, 35% of patients did not clinically improve after CRT. Objective reverse remodeling, typically defined as >15% reduction in the end-systolic volume, occurs in approximately 60% of patients. Most echocardiographic studies to date have reported only short- and intermediate-term results.

The objectives of the LOCATE-Pilot study are as follows: 1) to determine the proportion of patients undergoing CRT or CRT with defibrillator (CRT-D) with interpretable pulsed-wave tissue Doppler echocardiographic signals to quantitate and localize mechanical dyssynchrony; 2) to determine how frequently the LV lead can be successfully implanted in the most delayed basal segment (area of maximal delay); 3) to determine whether TDI guidance of CRT improves the proportion of patients with an echocardiographic response to treatment (reverse remodeling) at 6 months; 4) to determine whether TDI guidance of CRT improves the proportion of patients with a clinical response to treatment (6 min walk time, major clinical vascular events, or Minnesota Living with Heart Failure Quality of Life score); 5) to confirm that echocardiographic targeting of LV lead implantation is safe and does not hamper efficiency in the electrophysiological laboratory; 6) to validate the peak velocity delay (PVD) as a predictor of CRT response using pulsed-wave Doppler tissue imaging.

The LOCATE-pilot is a randomized, prospective study of 60 patients undergoing implantation of a Medtronic market approved CRT system. All patients will undergo a comprehensive baseline echocardiographic study in which a 6-segment model will be used to quantify dyssynchrony by the pulsed-wave Doppler technique. Myocardial viability will be assessed by conventional 2D criteria and nuclear perfusion data when available. Patients will be randomized to 1 of 2 groups with 30 patients per group on an intention-to-treat basis: 1) Control group: the implanting physician will have no knowledge of the baseline dyssynchrony assessment and use the current standard of care in the LV lead implantation; and 2) Echo-Guided group: the implanting physician will have full knowledge of baseline echocardiographic study and will use the dyssynchrony and viability data to guide final LV lead placement.

For this pilot study, patients will be followed for 6 months with a repeat Echocardiogram at 6 months. The primary endpoint of the study is indexed end systolic volume decrease >15% by biplane Simpson's technique.

ELIGIBILITY:
Inclusion Criteria:

* male/female patients
* NYHA class III and IV chronic heart failure
* symptoms refractory to standard therapy (beta blocker and either ACE-I or ARB on stable dosages for 1 month minimum and duration of 3 months therapy minimum)
* patient has signed and dated informed consent
* patient able to receive pectoral device implant
* QRS>= 130 ms
* EF <= 35%
* follow-up at Michigan Heart CHF clinic feasible
* patient understanding of protocol and willing to comply

Exclusion Criteria:

* recent myocardial infarction (<3 months)
* recent surgical or percutaneous revascularization (<3months)
* age < 18 months
* permanent AF without AV junction ablation
* life expectancy under 6 months
* women of child-bearing potential and not willing or able to take birth control
* mechanical tricuspid valve
* prior orthotopic heart transplantation
* intermittent inotropic therapy or inotropic-dependent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2007-04

PRIMARY OUTCOMES:
Efficacy: Indexed end systolic volume decrease>15% by biplane Simpson's technique at 6 month follow-up.
Safety: CRT implantation morbidity; mortality

SECONDARY OUTCOMES:
Clinical composite (6 month clinical assessment in HF clinic): 6 minute hall walk distance, MLWHF QOL score, NYHA functional classification
Clinical outcome at study termination (6 month follow-up for last patient enrolled): vital status (all cause mortality), cardiac mortality, unplanned hospitalization for major cardiovascular event
Proportion of diagnostic pulsed wave Doppler baseline studies
Success rate at Echo guided implantation (implantation of LV lead to target segment)
Outcomes stratified by concordance (pacing most delayed, viable segment)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Girard, MD, PhD, Principal Investigator — Michigan Heart, PC
Locations (1):
- Michigan Heart, PC, Ypsilanti, Michigan, United States

REFERENCES:
- [Background] McAlister FA, Ezekowitz JA, Wiebe N, Rowe B, Spooner C, Crumley E, Hartling L, Klassen T, Abraham W. Systematic review: cardiac resynchronization in patients with symptomatic heart failure. Ann Intern Med. 2004 Sep 7;141(5):381-90. doi: 10.7326/0003-4819-141-5-200409070-00101. Epub 2004 Aug 16. PMID 15353430
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Pitzalis MV, Iacoviello M, Romito R, Massari F, Rizzon B, Luzzi G, Guida P, Andriani A, Mastropasqua F, Rizzon P. Cardiac resynchronization therapy tailored by echocardiographic evaluation of ventricular asynchrony. J Am Coll Cardiol. 2002 Nov 6;40(9):1615-22. doi: 10.1016/s0735-1097(02)02337-9. PMID 12427414
- [Background] Bax JJ, Bleeker GB, Marwick TH, Molhoek SG, Boersma E, Steendijk P, van der Wall EE, Schalij MJ. Left ventricular dyssynchrony predicts response and prognosis after cardiac resynchronization therapy. J Am Coll Cardiol. 2004 Nov 2;44(9):1834-40. doi: 10.1016/j.jacc.2004.08.016. PMID 15519016
- [Background] Yu CM, Fung WH, Lin H, Zhang Q, Sanderson JE, Lau CP. Predictors of left ventricular reverse remodeling after cardiac resynchronization therapy for heart failure secondary to idiopathic dilated or ischemic cardiomyopathy. Am J Cardiol. 2003 Mar 15;91(6):684-8. doi: 10.1016/s0002-9149(02)03404-5. PMID 12633798
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368